CLINICAL TRIAL: NCT03226522
Title: A Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of AXS-05 for the Treatment of Agitation in Subjects With Dementia of the Alzheimer's Type
Brief Title: Addressing Dementia Via Agitation-Centered Evaluation
Acronym: ADVANCE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXS-05-AD-301
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type; Alzheimer Disease; Agitation,Psychomotor
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AXS-05 (Experimental): AXS-05 tablets taken by mouth for 5 weeks.
  Interventions: Drug: AXS-05
- Bupropion (Active Comparator): Bupropion tablets taken by mouth for 5 weeks.
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Placebo tablets taken by mouth for 5 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-05 — AXS-05
  Arms: AXS-05
Drug: Bupropion — Bupropion
  Arms: Bupropion
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study, to assess the efficacy and safety of AXS-05 in the treatment of agitation in patients with Alzheimer's disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) based on the 2011 National Institute on Aging-Alzheimer Association (NIA-AA) criteria.
* Diagnosis of clinically signification agitation resulting from probable AD according to the International Psychogeriatric Association (IPA) provisional definition of agitation.

Exclusion Criteria:

* Patient has dementia predominantly of non-Alzheimer's type.
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 366 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (72):
  - Axsome Study Site, Gilbert, Arizona
  - Axsome Study Site, Phoenix, Arizona
  - Axsome study site, Scottsdale, Arizona
  - Axsome Study Site, Tucson, Arizona
  - Axsome Study Site, Little Rock, Arkansas
  - Axsome study site, Canoga Park, California
  - Axsome study site, Costa Mesa, California
  - Axsome study site, Fresno, California
  - Axsome study site, Long Beach, California
  - Axsome Study Site, Los Alamitos, California
  - Axsome study site, Riverside, California
  - Axsome study site, Sacramento, California
  - Axsome study site, Santa Ana, California
  - Axsome Study Site, Santa Clarita, California
  - Axsome study site, Sherman Oaks, California
  - Axsome study site, Simi Valley, California
  - Axsome study site, Temecula, California
  - Axsome study site, Ventura, California
  - Axsome Study Site, Colorado Springs, Colorado
  - Axsome study site, Cromwell, Connecticut
  - Axsome study site, New London, Connecticut
  - Axsome Study Site, Apopka, Florida
  - Axsome study site, Boca Raton, Florida
  - Axsome study site, Boynton Beach, Florida
  - Axsome Study Site, Coconut Creek, Florida
  - Axsome Study Site, Greenacres City, Florida
  - Axsome study site, Hallandale, Florida
  - Axsome study site, Hialeah, Florida
  - Axsome Study Site, Lake City, Florida
  - Axsome study site, Miami, Florida
  - Axsome Study Site, Orlando, Florida
  - Axsome study site, Pensacola, Florida
  - Axsome Study Site, Port Orange, Florida
  - Axsome study site, Spring Hill, Florida
  - Axsome study site, Tampa, Florida
  - Axsome study site, Atlanta, Georgia
  - Axsome study site, Decatur, Georgia
  - Axsome Study Site, Honolulu, Hawaii
  - Axsome study site, Boise, Idaho
  - Axsome Study Site, Flossmoor, Illinois
  - Axsome study site, Avon, Indiana
  - Axsome Study Site, Overland Park, Kansas
  - Axsome Study Site, Topeka, Kansas
  - Axsome study site, Baton Rouge, Louisiana
  - Axsome Study Site, Lake Charles, Louisiana
  - Axsome Study Site, Hattiesburg, Mississippi
  - Axsome study site, Chesterfield, Missouri
  - Axsome Study Site, St Louis, Missouri
  - Axsome study site, Las Vegas, Nevada
  - Axsome Study Site, Las Vegas, Nevada
  - Axsome Study Site, Princeton, New Jersey
  - Axsome study site, Toms River, New Jersey
  - Axsome Study Site, Albany, New York
  - Axsome study site, Brooklyn, New York
  - Axsome study site, New York, New York
  - Axsome study site, Staten Island, New York
  - Axsome Study Site, Charlotte, North Carolina
  - Axsome study site, Charlotte, North Carolina
  - Axsome Study Site, Winston-Salem, North Carolina
  - Axsome study site, Cincinnati, Ohio
  - Axsome Study Site, Dayton, Ohio
  - Axsome study site, Shaker Heights, Ohio
  - Axsome Study Site, Oklahoma City, Oklahoma
  - Axsome study site, DeSoto, Texas
  - Axsome Study Site, McKinney, Texas
  - Axsome study site, Wichita Falls, Texas
  - Axsome study site, Orem, Utah
  - Axsome Study Site, Charlottesville, Virginia
  - Axsome Study Site, Richmond, Virginia
  - Axsome study site, Bellevue, Washington
  - Axsome Study Site, Everett, Washington
  - Axsome study site, Spokane, Washington
- Axsome study site, Caulfield, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Groups:
- AXS-05: AXS-05 tablets taken twice daily for 5 weeks.
  AXS-05: AXS-05
- Bupropion: Bupropion tablets taken twice daily for 5 weeks.
  Bupropion: Bupropion
- Placebo: Placebo tablets taken twice daily for 5 weeks.
  Placebo: Placebo
Period: Overall Study
Arm/Group | AXS-05 | Bupropion | Placebo
Started | 159 | 49 | 158
Safety Population | 159 | 49 | 158
mITT Population | 152 | 49 | 156
Completed | 137 | 48 | 136
Not Completed | 22 | 1 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AXS-05 | Bupropion | Placebo | Total
Number analyzed (Participants) | 159 | 49 | 158 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (5.71) | 76.4 (6.13) | 74.6 (6.11) | 75.1 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 22 | 92 | 205
  Male | 68 | 27 | 66 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 0 | 0 | 2
  Race: Asian | 2 | 0 | 1 | 3
  Race: Black or African American | 12 | 5 | 25 | 42
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Race: Other | 1 | 1 | 0 | 2
  Race: Unknown or Not Reported | 1 | 0 | 1 | 2
  Race: White | 141 | 43 | 130 | 314

OUTCOME MEASURES:

1. Primary Outcome: Change in CMAI Total Score
Description: The Cohen-Mansfield Agitation Inventory (CMAI) is a 29-item caregiver-rated questionnaire that assesses the frequency of agitation-related and disruptive behaviors in subjects with dementia. The scale contains 29 behaviors or items organized into four subscales: physically aggressive, physically non-aggressive, verbally aggressive, and verbally non-aggressive. The CMAI is administered by interviewing the caregiver and asking him or her to rate the frequency with which the subject manifests each behavior using a seven-point scale: 1=never (better outcome), 7=several times an hour (worse outcome). The CMAI total score is the sum of the scores for all of the items in the CMAI. CMAI total scores range from a minimum of 29 (better outcome) to a maximum of 203 (worse outcome).
Time Frame: 5 weeks
Population: modified Intent-to-Treat (mITT) Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AXS-05 | Bupropion | Placebo
Number analyzed (Participants) | 152 | 49 | 156
score on a scale | -15.4 (1.25) | -10.0 (3.02) | -11.5 (1.10)
Statistical Analysis 1: Comparison: AXS-05 vs Placebo; Test type: Superiority; p = 0.010, Mixed Models Analysis
Statistical Analysis 2: Comparison: AXS-05 vs Bupropion; Test type: Superiority; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the Baseline visit through 30 days after the last study visit (up to 10 weeks).
Description: Safety Population
Arm/Group | AXS-05 | Bupropion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/159 | 1/49 | 1/158
Serious Adverse Events (participants affected / at risk) | 5/159 | 4/49 | 9/158
Other Adverse Events (participants affected / at risk) | 33/159 | 17/49 | 24/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=159) | Bupropion (N=49) | Placebo (N=158)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=159) | Bupropion (N=49) | Placebo (N=158)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 3 (4) | 7 (7)
Fatigue (General disorders) | 3 (3) | 5 (5) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 4 (13) | 7 (11) | 3 (3)
Dizziness (Nervous system disorders) | 10 (11) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 6 (8) | 3 (3) | 4 (5)
Somnolence (Nervous system disorders) | 13 (13) | 2 (2) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (2) | 3 (3) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT03226522/Prot_SAP_000.pdf